CLINICAL TRIAL: NCT04604275
Title: Functional Sucrase Deficiency in Short Bowel Syndrome Patients With Intestinal Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to recruit further patients for study
Sponsor: University of Miami (Other)
Collaborators: QOL Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20191253
Record Dates: First submitted 2020-10-22; First posted 2020-10-27 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Short Gut Syndrome
Keywords: Intestinal failure
MeSH Terms: conditions — Short Bowel Syndrome; Intestinal Failure | interventions — Sucrase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sucrase intervention followed by placebo (Experimental): Participants in this arm will receive sucrase for 4 weeks followed by wash out of 1 week with no drug administered then 4 weeks of placebo.
  Interventions: Drug: Sucrase; Other: Placebo
- Placebo followed by sucrase intervention (Experimental): Participants in this arm will receive placebo for 4 weeks followed by wash out of 1 week with no drug administered then 4 weeks of sucrase.
  Interventions: Drug: Sucrase; Other: Placebo

INTERVENTIONS:
Drug: Sucrase — 1 mL (8,500 I.U.) (one full measuring scoop or 28 drops) per meal or snack for patients up to 15 kg in body weight. 2 mL (17,000 I.U.) for patients over 15kg in body weight. Dosage is 1 or 2 mL (8,500 to 17,000 I.U.) taken orally or by g-tube with each meal or snack diluted in water, milk, or infant formula.
Other: Placebo — 1 mL of placebo per meal or snack for patients up to 15 kg in body weight. 2 mL of placebo per meal of snack for patients above 15kg in body weight. Dosage is 1 or 2 mL of placebo taken orally or by g-tube with each meal or snack diluted in water, milk, or infant formula.

SUMMARY:
Short gut syndrome with intestinal failure patients may have decreased production of disaccharidases, like sucrase, an enzyme responsible for digesting sugar in foods. This can happen due to loss of bowel length from surgery or from loss of cellular function in the intestines due to use of parenteral nutrition intravenously. Therefore, patients with these conditions may not be able to digest sucrose (sugar) fully. Patients might experience abdominal distension/pain, vomiting and diarrhea when sugar is taken in orally or through the g-tube, which can limit patients' ability to increase oral or g-tube feeds in short gut syndrome patients with intestinal failure.

In patients with short gut syndrome and intestinal failure, the administration of exogenous sucrase (enzyme) may improve sucrose (sugar) digestion and thus the ability to tolerate more oral or g-tube feeds.

ELIGIBILITY:
Inclusion Criteria:

* Short bowel syndrome, of all ages, with dependence on parental support to provide at least 50% of fluid or caloric needs.
* Must be on diet containing sucrose.
* Must be willing and able to sign informed consent
* Adult and Pediatric patients (all ages)

Exclusion Criteria:

* Current IV antibiotic administration for confirmed bout of bacteremia.
* No enteral nutrition
* Any condition, disease, illness, or circumstance that in the investigator's opinion puts the subject at any undue risk, prevents completion of the study, or interferes with analysis of the study results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Fifi, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Intervention 1
Arm/Group | Sucrase Intervention Followed by Placebo | Placebo Followed by Sucrase Intervention
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0
Period: Washout-1 Week
Arm/Group | Sucrase Intervention Followed by Placebo | Placebo Followed by Sucrase Intervention
Started | 2 | 1
Completed | 1 | 1
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Intervention 2
Arm/Group | Sucrase Intervention Followed by Placebo | Placebo Followed by Sucrase Intervention
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sucrase Intervention Followed by Placebo | Placebo Followed by Sucrase Intervention | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Carbohydrate Malabsorption
Description: Degree of carbohydrate malabsorption will be assessed by decrease in number of stools per day.
Time Frame: baseline, 9 weeks
Population: Due to operational challenges across multiple study sites, the required data for this outcome measure could not be collected or retained. The study involved several coordinators working across dispersed locations, which introduced variability in data handling and documentation practices. Although standardized procedures were in place, inconsistencies emerged in how forms were distributed, tracked, and returned.
Arm/Group | Sucrase Intervention Followed by Placebo | Placebo Followed by Sucrase Intervention
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Carbohydrate Malabsorption as Measured by Patient Symptom Survey
Description: Degree of carbohydrate malabsorption will be assessed by change in patient symptomatology by change in score on patient symptom survey.
  The survey has range from 0-52 with higher score being worse symptoms and lower being better.
Time Frame: baseline, 9 weeks
Population: as for outcome 1
Arm/Group | Sucrase Intervention Followed by Placebo | Placebo Followed by Sucrase Intervention
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Carbohydrate Malabsorption as Measured by Growth Velocity
Description: Carbohydrate malabsorption will be measured by increase in growth velocity in kg/week
Time Frame: baseline, 9 weeks
Population: as for outcome 1
Arm/Group | Sucrase Intervention Followed by Placebo | Placebo Followed by Sucrase Intervention
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change in Carbohydrate Malabsorption as Measured by Enteral Nutrition Tolerance
Description: Carbohydrate malabsorption will be measured by ability to advance enteral nutrition in ml/day
Time Frame: baseline, 9 weeks
Population: as for outcome 1
Arm/Group | Sucrase Intervention Followed by Placebo | Placebo Followed by Sucrase Intervention
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Digestion
Description: Change in digestion will be measured by change in abdominal distension/girth measured in cm
Time Frame: baseline, 9 weeks
Population: as for outcome 1
Arm/Group | Sucrase Intervention Followed by Placebo | Placebo Followed by Sucrase Intervention
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Digestion as Measured by Amount of Emesis
Description: Change in digestion will be assessed by number of emesis per day
Time Frame: baseline, 9 weeks
Population: as for outcome 1
Arm/Group | Sucrase Intervention Followed by Placebo | Placebo Followed by Sucrase Intervention
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Digestion as Measured by Stool Consistency
Description: Change in digestion will be assessed as a change in stool consistency from liquid (7) to solid(1) using Bristol stool chart
Time Frame: baseline, 9 weeks
Population: as for outcome 1
Arm/Group | Sucrase Intervention Followed by Placebo | Placebo Followed by Sucrase Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 weeks
Description: Adverse Events are being reported per arm. There are only 2 arms for this study.
Arm/Group | Sucrase Intervention Followed by Placebo | Placebo Followed by Sucrase Intervention
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

LIMITATIONS AND CAVEATS:
The study was terminated due to low accrual. The target population consisted of individuals with a rare condition that is not commonly found in the general population, which significantly limited recruitment feasibility. Despite outreach efforts and engagement with specialized clinical sites, the rarity of the condition and strict eligibility criteria resulted in insufficient enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT04604275/Prot_000.pdf